CLINICAL TRIAL: NCT05983796
Title: Prospective Study of 18F-HER2 PET in Evaluating the Efficacy of Anti-HER2 Therapy for Urothelial Carcinoma.
Brief Title: 18F-HER2 PET in Evaluating the Efficacy of Anti-HER2 Therapy for Urothelial Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIT20230066C
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: 18F-HER2 PET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-HER2 PET (Experimental)
  Interventions: Diagnostic Test: 18F-HER2 PET

INTERVENTIONS:
Diagnostic Test: 18F-HER2 PET — 18F-HER2 PET

SUMMARY:
This is a open-label, one-arm, multicenter study aimed to explore the efficacy and safety of 18F-HER2 PET in Evaluating the Efficacy of Anti-HER2 Therapy for Urothelial Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent document must be signed.
2. Aged 30-80 years old, both genders.
3. Patients with locally advanced or advanced urothelial carcinoma
4. Patients plan to undergo anti HER2 treatment.

Exclusion Criteria:

1. Subjects with active malignancies other than urothelial carcinoma within 5 years should be excluded.
2. Patients with severe liver, kidney, and hematopoietic diseases
3. Patients with other mental disorders or primary emotional disorders
4. Those who are unable to understand, comply with the research protocol, or sign an informed consent form
5. PET imaging Contraindication (including pregnant women, lactating women, women of childbearing age who have a recent fertility plan, etc.)
6. Individuals who are allergic to imaging agents
7. Hypoglycemic reactions, severe pain, etc. cannot be accompanied by PET scans

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the Efficacy of Anti-HER2 Therapy for Urothelial Carcinoma | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhen Shan, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No